CLINICAL TRIAL: NCT04041700
Title: A Prospective, Multicentre, Open Clinical Investigation Evaluating Clinical Performance, Safety and Patient Reported Outcomes With an Active Osseointegrated Steady-State Implant System (OSI) in Adult Subjects With Conductive Hearing Loss, Mixed Hearing Loss or Single-sided Sensorineural Deafness
Brief Title: Clinical Performance, Safety and Patient Reported Outcomes of an Active Osseointegrated Steady-State Implant System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Statistiska Konsultgruppen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBAS5751
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss
Keywords: Hearing Loss, Conductive; Hearing Loss, Mixed; Deafness, sensorineural single-sided
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osia 2 system (Experimental)
  Interventions: Device: Osia 2 system

INTERVENTIONS:
Device: Osia 2 system — System includes the OSI200 implant surgically placed under the skin behind the ear, the BI300 implant osseointegrated in the bone and the external Osia 2 sound processor.

SUMMARY:
The aim of this clinical investigation is to collect data on objective and subjective hearing performance, quality of life and safety in adult subjects with conductive hearing loss, mixed hearing loss or single-sided sensorineural deafness.

ELIGIBILITY:
Inclusion Criteria:

* Subject with conductive hearing loss or mixed hearing loss in the ear to be implanted. Bone conduction thresholds with pure tone average (PTA4; mean of 0.5, 1, 2 and 4 kHz) of ≤ 55 dB sensorineural hearing loss.

OR Subject with single-sided sensorineural deafness who is a candidate for Baha surgery. Air conduction thresholds with a pure tone average PTA4 (mean of 0.5, 1, 2 and 3 kHz) of ≤ 20 dB sensorineural hearing loss in the good ear OR subject who is indicated for an (Air Conduction-Contralateral Routing of Signal (AC CROS) but-for some reason-cannot or will not use an AC CROS.

* Adult subjects (18 years or older).
* Previous experience from amplified sound through properly fitted amplification (for example but not limited to Hearing aid, Contralateral Routing of Signal (CROS) device, Bone conduction hearing device on softband).
* Candidate is a fluent speaker in the language used to assess speech perception performance.
* Willing and able to provide written informed consent

Exclusion Criteria:

* Uncontrolled diabetes as judged by the investigator.
* Condition that could jeopardise osseointegration and/or wound healing (e.g. osteoporosis, psoriasis, long-term systemic use of corticosteroids) or condition that may have an impact on the outcome of the investigation as judged by the investigator.
* Insufficient bone quality and quantity to support successful implant placement.
* Previous surgery and/or implantation with any bone conduction/active device on the side to be implanted, which may jeopardise the implantation and use of the Osia 2 system, as judged by the investigator.
* Use of ototoxic drugs that could be harmful to the hearing, as judged by the investigator.
* Unable to follow investigational procedures, e.g. to complete quality of life scales, or unwilling to comply with the requirements of the clinical investigation as determined by the investigator.
* Condition with a likely negative progression and/or with expected relapses jeopardising general wellbeing and health-related quality of life as judged by the investigator.
* Subject that has received radiotherapy in the area of implantation or is planned for such radiotherapy during the study period.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation
* Currently participating, or participated within the last 30 days, in another interventional clinical investigation involving an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Ganlöv, Study Director — Cochlear
Locations (3):
- Australia (2):
  - Sydney Cochlear Implant Centre, Gladesville
  - The Royal Victorian Eye and Ear Hospital, Melbourne
- Department of Otorhinolaryngology, Head and Neck Surgery Faculty of Medicine. The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cowan R, Lewis AT, Hallberg C, Tong MCF, Birman CS, Ng IH, Briggs R. Clinical performance, safety, and patient-reported outcomes of an active osseointegrated bone-conduction hearing implant system at 24-month follow-up. Eur Arch Otorhinolaryngol. 2024 Feb;281(2):683-691. doi: 10.1007/s00405-023-08133-3. Epub 2023 Aug 8. PMID 37552281
- [Derived] Briggs R, Birman CS, Baulderstone N, Lewis AT, Ng IHY, Ostblom A, Rousset A, Tari S, Tong MCF, Cowan R. Clinical Performance, Safety, and Patient-Reported Outcomes of an Active Osseointegrated Steady-State Implant System. Otol Neurotol. 2022 Aug 1;43(7):827-834. doi: 10.1097/MAO.0000000000003590. PMID 35878640

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 participants were recruited in three centres from 16 August 2019 to 24 September 2020.
Period: Overall Study
Arm/Group | Osia 2 System
Started | 29
Completed | 27
Not Completed | 2
Not completed — Pregnancy | 1
Not completed — Unable to visit the site due to the Covid-19 travel restrictions | 1

BASELINE CHARACTERISTICS:
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Hong Kong | 3
  Australia | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Hearing Performance With the Osia 2 System at 3 Months Post-surgery Compared to Preoperative Unaided Condition Assessed Via Audiometric Thresholds
Description: Free field (Pure Tone Average 4, mean of 0.5, 1,2 and 4 kHz)
Time Frame: Baseline before surgery, 3 months after surgery
Population: Data was only received for 27 participants. One participant did not receive the sound processor due to the Covid-19 pandemic and one participant did not attend neither the 4 weeks visit nor the 3 months visit.
Measure: Mean (Standard Deviation); unit: db HL (decibel Hearing Level)
Arm/Group | Osia 2 System
Number analyzed (Participants) | 27
db HL (decibel Hearing Level) | -27.3 (8.7)

2. Primary Outcome: Change in Hearing Performance With the Osia 2 System at 3 Months Post-surgery Compared to Preoperative Unaided Situation Assessed Via Adaptive Speech Recognition in Noise
Description: Speech-to-noise ratio, 50% speech understanding
Time Frame: Baseline before surgery, 3 months after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: db SNR (decibel Speech in Noise Ratio)
Arm/Group | Osia 2 System
Number analyzed (Participants) | 27
db SNR (decibel Speech in Noise Ratio) | -9.10 (7.88)

3. Secondary Outcome: Change in Hearing Performance With the Osia 2 System at 4 Weeks and 6 Months Post Surgery Compared to Preoperative Unaided Situation Assessed Via Audiometric Thresholds
Description: Free field (Pure Tone Average 4, mean of 0.5, 1,2 and 4 kHz)
Time Frame: Baseline before surgery, 4 weeks and 6 months after surgery
Population: At 4 weeks, data was only received for 27 participants. One participant did not receive the sound processor due to the Covid-19 pandemic and one participant did not attend neither the 4 weeks visit nor the 3 months visit.
  At 6 months visit, data was received for 28 participants.The participant that did not attend previous visits did visit the site and data was collected. The participant that did not receive the sound processor still could not visit site.
Measure: Mean (Standard Deviation); unit: db HL (decibel Hearing Level)
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
db HL (decibel Hearing Level)
  4 weeks: number analyzed (Participants) | 27
  4 weeks | -25.6 (8.3)
  6 months | -28.4 (9.6)

4. Secondary Outcome: Change in Hearing Performance With the Osia 2 System at 4 Weeks and 6 Months Post Surgery Compared to Preoperative Unaided Situation Assessed Via Adaptive Speech Recognition in Noise
Description: Speech-to-noise ratio, 50% speech understanding
Time Frame: Baseline before surgery, 4 weeks and 6 months after surgery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: db SNR (decibel Speech in Noise Ratio)
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
db SNR (decibel Speech in Noise Ratio)
  4 weeks: number analyzed (Participants) | 27
  4 weeks | -8.76 (8.06)
  6 months | -8.84 (7.88)

5. Secondary Outcome: Change in Hearing Performance With the Osia 2 System at 4 Weeks, 3 Months and 6 Months Post Surgery Compared to Preoperative Unaided Situation Assessed Via Audiometric Thresholds
Description: Free-field [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 and 8.0 kHz]
Time Frame: Baseline before surgery, 4 weeks, 3 months and 6 months after surgery
Population: At the 4 weeks and 3 months visits, data was only received for 27 participants. One participant did not receive the sound processor due to the Covid-19 pandemic and one participant did not attend neither the 4 weeks visit nor the 3 months visit.
  At the 6 months visit, data was received for 28 participants. The participant that did not attend previous visits did visit the site and data was collected. The participant that did not receive the sound processor still could not visit site.
Measure: Mean (Standard Deviation); unit: db HL (decibel Hearing Level)
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
db HL (decibel Hearing Level)
  0.25 kHz, 4 weeks: number analyzed (Participants) | 27
  0.25 kHz, 4 weeks | -13.5 (12.0)
  0.5 kHz, 4 weeks: number analyzed (Participants) | 27
  0.5 kHz, 4 weeks | -23.1 (12.1)
  0.75 kHz, 4 weeks: number analyzed (Participants) | 27
  0.75 kHz, 4 weeks | -30.2 (10.6)
  1.0 kHz, 4 weeks: number analyzed (Participants) | 27
  1.0 kHz, 4 weeks | -28.3 (10.1)
  1.5 kHz, 4 weeks: number analyzed (Participants) | 27
  1.5 kHz, 4 weeks | -30.0 (10.7)
  2.0 kHz, 4 weeks: number analyzed (Participants) | 27
  2.0 kHz, 4 weeks | -25.7 (9.7)
  3.0 kHz, 4 weeks: number analyzed (Participants) | 27
  3.0 kHz, 4 weeks | -24.8 (11.6)
  4.0 kHz, 4 weeks: number analyzed (Participants) | 27
  4.0 kHz, 4 weeks | -25.4 (11.3)
  6.0 kHz, 4 weeks: number analyzed (Participants) | 27
  6.0 kHz, 4 weeks | -35.0 (11.9)
  8.0 kHz, 4 weeks: number analyzed (Participants) | 27
  8.0 kHz, 4 weeks | -5.44 (12.9)
  0.25 kHz, 3 months: number analyzed (Participants) | 27
  0.25 kHz, 3 months | -14.8 (11.1)
  0.5 kHz, 3 months: number analyzed (Participants) | 27
  0.5 kHz, 3 months | -24.4 (11.2)
  0.75 kHz, 3 months: number analyzed (Participants) | 27
  0.75 kHz, 3 months | -32.0 (10.8)
  1.0 kHz, 3 months: number analyzed (Participants) | 27
  1.0 kHz, 3 months | -29.1 (10.2)
  1.5 kHz, 3 months: number analyzed (Participants) | 27
  1.5 kHz, 3 months | -30.6 (11.3)
  2.0 kHz, 3 months: number analyzed (Participants) | 27
  2.0 kHz, 3 months | -27.0 (10.9)
  3.0 kHz, 3 months: number analyzed (Participants) | 27
  3.0 kHz, 3 months | -25.2 (11.5)
  4.0 kHz, 3 months: number analyzed (Participants) | 27
  4.0 kHz, 3 months | -28.7 (11.5)
  6.0 kHz, 3 months: number analyzed (Participants) | 27
  6.0 kHz, 3 months | -36.5 (12.1)
  8.0 kHz, 3 months: number analyzed (Participants) | 27
  8.0 kHz, 3 months | -8.59 (13.8)
  0.25 kHz, 6 months | -14.3 (12.8)
  0.5 kHz, 6 months | -24.6 (12.2)
  0.75 kHz, 6 months | -32.0 (11.5)
  1.0 kHz, 6 months | -31.3 (11.1)
  1.5 kHz, 6 months | -33.8 (10.9)
  2.0 kHz, 6 months | -28.4 (12.3)
  3.0 kHz, 6 months | -26.6 (9.9)
  4.0 kHz, 6 months | -29.3 (11.3)
  6.0 kHz, 6 months | -37.3 (12.5)
  8.0 kHz, 6 months | -7.71 (15.9)

6. Secondary Outcome: Change in Hearing Performance With the Osia 2 System at 4 Weeks, 3 Months and 6 Months Post Surgery Compared to Preoperative Unaided Situation Assessed Via Speech Recognition in Quiet
Description: % correctly perceived words at 50dB, 65dB and 80dB SPL
Time Frame: Baseline before surgery, 4 weeks, 3 months and 6 months after surgery
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of correct words
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
Percentage of correct words
  Speech in quiet at 50 dB, 4 weeks: number analyzed (Participants) | 27
  Speech in quiet at 50 dB, 4 weeks | 62.7 (20.7)
  Speech in quiet at 65 dB, 4 weeks: number analyzed (Participants) | 27
  Speech in quiet at 65 dB, 4 weeks | 55.1 (29.4)
  Speech in quiet at 80 dB, 4 weeks: number analyzed (Participants) | 27
  Speech in quiet at 80 dB, 4 weeks | 23.9 (27.5)
  Speech in quiet at 50 dB, 3 months: number analyzed (Participants) | 27
  Speech in quiet at 50 dB, 3 months | 63.8 (21.6)
  Speech in quiet at 65 dB, 3 months: number analyzed (Participants) | 27
  Speech in quiet at 65 dB, 3 months | 55.5 (29.3)
  Speech in quiet at 80 dB, 3 months: number analyzed (Participants) | 27
  Speech in quiet at 80 dB, 3 months | 23.7 (27.7)
  Speech in quiet at 50 dB, 6 months | 62.3 (22.1)
  Speech in quiet at 65 dB, 6 months | 54.0 (29.8)
  Speech in quiet at 80 dB, 6 months | 24.3 (28.0)

7. Secondary Outcome: Change in Self-reported Hearing Outcome With the Osia 2 System at 3 Months and 6 Months Post Surgery Compared to the Preoperative Unaided Situation Via Abbreviated Profile of Hearing Aid Benefit (APHAB) Questionnaire
Description: Measuring change of Ease of communication, Reverberation, Background noise, Aversiveness and a Global score with the Osia 2 System from the pre-operative unaided situation. The absolute APHAB scale is between 0 and 100%, where 0% indicates no problems and 100% indicates always problem. The change from unaided to aided hearing is presented. A positive value indicates an impairment, a negative value an improvement.
Time Frame: Baseline before surgery, 3 months and 6 months after surgery
Population: One participant did not receive the sound processor and did not perform this questionnaire at either 3- or 6-months visit.
  One participant did not perform this questionnaire at 3-month visit and another participant did not perform this questionnaire at the 6-month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osia 2 System
Number analyzed (Participants) | 27
units on a scale
  APHAB - Ease of communication, 3 months | 28.1 (30.7)
  APHAB - Background Noise, 3 months | 27.6 (26.9)
  APHAB - Reverberation, 3 months | 20.3 (24.3)
  APHAB - Aversiveness, 3 months | -5.2 (34.9)
  APHAB - Global, 3 months | 25.4 (25.0)
  APHAB - Ease of communication, 6 months | 27.4 (31.4)
  APHAB - Background Noise, 6 months | 28.7 (28.1)
  APHAB - Reverberation, 6 months | 21.7 (26.4)
  APHAB - Aversiveness, 6 months | -0.212 (33.0)
  APHAB - Global, 6 months | 25.9 (26.2)

8. Secondary Outcome: Change in Self-reported Hearing Outcome With the Osia 2 System at 3 Months and 6 Months Post Surgery Compared to the Preoperative Unaided Situation Via the Speech, Spatial and Qualities of Hearing Scale (SSQ) Questionnaire
Description: Measuring change of speech, spatial and hearing experiences with the Osia 2 System from the pe-operative unaided situation. A scale from 0 to 10 is used, where 0 represents "can not hear at all", and 10 "hear perfectly". The change from unaided to aided hearing is presented. A positive value indicates improved hearing, a negative value indicates impaired hearing.
Time Frame: Baseline before surgery, 3 months and 6 months after surgery
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Osia 2 System
Number analyzed (Participants) | 27
Score on a scale
  SSQ12 Total score, 3 months | 2.88 (1.56)
  SSQ12 Speech score, 3 months | 3.12 (1.78)
  SSQ12 Spatial score, 3 months | 2.92 (2.07)
  SSQ12 Quality score, 3 months | 2.55 (1.78)
  SSQ12 Total score, 6 months | 2.50 (1.66)
  SSQ12 Speech score, 6 months | 2.68 (1.89)
  SSQ12 Spatial score, 6 months | 2.30 (2.42)
  SSQ12 Quality score, 6 months | 2.41 (1.81)

9. Secondary Outcome: Change in Health-related Quality of Life With the Osia 2 System at 3 Months and 6 Months Post Surgery Compared to the Preoperative Unaided Situation Via the Health Utilities Index Mark III (HUI) Questionnaire
Description: Change of health status and health related quality of life using the generic quality of life scale Health Utilities Index (HUI3) when wearing Osia 2 System compared to the pre-operative unaided situation. A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. The change from unaided to aided hearing is presented. A positive value indicates an improved quality of life, a negative value indicates impaired quality of life.
Time Frame: Baseline before surgery, 3 months and 6 months after surgery
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Osia 2 System
Number analyzed (Participants) | 27
score on a scale
  Comprehensive Health State, 3 months | 0.097 (0.167)
  Vision attribute, 3 months | 0.002 (0.017)
  Hearing attribute, 3 months | 0.113 (0.288)
  Speech attribute, 3 months | 0.006 (0.076)
  Ambulation attribute, 3 months | -0.006 (0.033)
  Dexterity attribute, 3 months | 0.031 (0.117)
  Emotion attribute, 3 months | 0.033 (0.071)
  Cognition attribute, 3 months | 0.011 (0.040)
  Pain attribute (HUI3), 3 months | 0.009 (0.061)
  Comprehensive Health State, 6 months | 0.091 (0.165)
  Vision attribute, 6 months | -0.004 (0.013)
  Hearing attribute, 6 months | 0.129 (0.318)
  Speech attribute, 6 months | 0.000 (0.106)
  Ambulation attribute, 6 months | 0.013 (0.045)
  Dexterity attribute, 6 months | 0.026 (0.120)
  Emotion attribute, 6 months | 0.020 (0.063)
  Cognition attribute, 6 months | 0.001 (0.064)
  Pain attribute (HUI3), 6 months | 0.011 (0.123)

10. Secondary Outcome: Surgical Information: Soft Tissue Thickness
Description: Measured in mm
Time Frame: Baseline before surgery or at surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
mm | 6.62 (1.29)

11. Secondary Outcome: Surgical Information: Surgery Time
Description: Time in minutes between first incision to last suture
Time Frame: At surgery
Population: Surgery time was not measured for one of the participants.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
min | 52.8 (13.3)

12. Secondary Outcome: Surgical Information: Bone Polishing/Removal at the Actuator Site
Description: Yes/No
Time Frame: At surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
Participants
  Yes | 12
  No | 17

13. Secondary Outcome: Surgical Information: BI300 Implant Length
Description: 3 mm/4 mm
Time Frame: At surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
Participants
  3 mm | 0
  4 mm | 29

14. Secondary Outcome: Surgical Information: Location of BI300 Implant
Description: Measured in mm between the ear canal and the center of the actuator
Time Frame: At surgery
Population: Data only gathered for 26 participants.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Osia 2 System
Number analyzed (Participants) | 26
mm | 52.9 (7.3)

15. Secondary Outcome: Surgical Information: Type of Anesthesia
Description: General/local
Time Frame: At surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
Participants
  General | 29
  Local | 0

16. Secondary Outcome: Surgical Information: Soft Tissue Reduction
Description: Yes/No
Time Frame: At surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
Participants
  Yes | 0
  No | 29

17. Secondary Outcome: Surgical Information: Surgical Incision Type
Description: Examples: C-shaped/S-shaped/straight
Time Frame: At surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
Participants
  C-shaped | 12
  S-shaped | 12
  Other | 5
  Straight | 0

18. Secondary Outcome: Surgical Information: Location of the Surgical Incision in Relation to the Actuator
Description: Anterior/posterior
Time Frame: At surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
Participants
  Anterior | 26
  Posterior | 3

19. Secondary Outcome: Surgical Information: Estimated Length of the Surgical Incision
Description: Measured in mm
Time Frame: At surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
mm | 71.4 (23.1)

20. Secondary Outcome: Surgical Information: Placement of the Coil
Description: Periosteal pocket (under periosteal)/on top of periosteum/on top of muscle)
Time Frame: At surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Osia 2 System
Number analyzed (Participants) | 29
Participants
  Periosteal pocket (under periosteal) | 24
  on top of periosteum | 3
  on top of muscle | 2

21. Secondary Outcome: Usability Information: Magnet Choice
Description: Magnet strength ranging from 1 to 4 where 1 is the weakest and 4 the strongest. A magnet allows the external sound processor to be placed in the correct position over the implanted system including an internal magnet.
Time Frame: At 4 weeks, 6 weeks, 3 months and 6 months after surgery
Population: For some participants the data are not available at all visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
Participants
  Magnet strength 2, 4 weeks | 1
  Magnet strength 3, 4 weeks | 11
  Magnet strength 4, 4 weeks | 16
  Magnet strength 2, 6 weeks: number analyzed (Participants) | 27
  Magnet strength 2, 6 weeks | 1
  Magnet strength 3, 6 weeks: number analyzed (Participants) | 27
  Magnet strength 3, 6 weeks | 13
  Magnet strength 4, 6 weeks: number analyzed (Participants) | 27
  Magnet strength 4, 6 weeks | 13
  Magnet strength 2, 3 months | 4
  Magnet strength 3, 3 months | 10
  Magnet strength 4, 3 months | 14
  Magnet strength 2, 6 months: number analyzed (Participants) | 27
  Magnet strength 2, 6 months | 4
  Magnet strength 3, 6 months: number analyzed (Participants) | 27
  Magnet strength 3, 6 months | 12
  Magnet strength 4, 6 months: number analyzed (Participants) | 27
  Magnet strength 4, 6 months | 11

22. Secondary Outcome: Usability Information: Sound Processor Retention
Description: Assessed via a Visual Analog Scale 100 mm where 0 mm represents insufficient retention and 100 mm excellent retention
Time Frame: At 4 weeks, 6 weeks, 3 months and 6 months after surgery
Population: Some participants did not perform the test at all visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osia 2 System
Number analyzed (Participants) | 27
units on a scale
  Overall Retention, 4 weeks: number analyzed (Participants) | 25
  Overall Retention, 4 weeks | 72.1 (22.8)
  Overall Retention, 6 weeks | 86.9 (13.9)
  Overall Retention, 3 months | 80.4 (17.1)
  Overall Retention, 6 months | 71.4 (26.7)

23. Secondary Outcome: Usability Information: Sound Processor Wearing Comfort
Description: Assessed via a Visual Analog Scale 100 mm where 0 mm represents no comfort at all and 100 mm excellent comfort
Time Frame: At 4 weeks, 6 weeks, 3 months and 6 months after surgery
Population: Some participants did not perform the test at all visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Osia 2 System
Number analyzed (Participants) | 27
units on a scale
  Overall Comfort, 4 weeks: number analyzed (Participants) | 25
  Overall Comfort, 4 weeks | 81.7 (14.1)
  Overall Comfort, 6 weeks | 87.1 (16.8)
  Overall Comfort, 3 months | 83.5 (16.4)
  Overall Comfort, 6 months | 81.4 (20.0)

24. Secondary Outcome: Usability Information: Use of SoftWear Pad
Description: Yes/No
Time Frame: At 6 weeks, 3 months and 6 months after surgery
Population: For some participants the data are not available at all visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
Participants
  Yes, 6 weeks: number analyzed (Participants) | 27
  Yes, 6 weeks | 3
  No, 6 weeks: number analyzed (Participants) | 27
  No, 6 weeks | 24
  Yes, 3 months | 4
  No, 3 months | 24
  Yes, 6 months: number analyzed (Participants) | 27
  Yes, 6 months | 2
  No, 6 months: number analyzed (Participants) | 27
  No, 6 months | 25

25. Secondary Outcome: Usability Information: Daily Use of Sound Processor
Description: Average hours of daily use
Time Frame: At 6 weeks, 3 months and 6 months after surgery
Population: For some participants the data are not available at all visits.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
hours/day
  Daily use, 6 weeks: number analyzed (Participants) | 27
  Daily use, 6 weeks | 10.3 (4.4)
  Daily use, 3 months | 9.57 (4.19)
  Daily use, 6 months: number analyzed (Participants) | 26
  Daily use, 6 months | 8.63 (4.67)

26. Secondary Outcome: Usability Information: Daily Streaming Time of Sound Processor
Description: Average hours of daily streaming
Time Frame: At 6 weeks, 3 months and 6 months after surgery
Population: For some participants the data are not available at all visits.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
hours/day
  Streaming, 6 weeks: number analyzed (Participants) | 27
  Streaming, 6 weeks | 0.407 (0.931)
  Streaming, 3 months | 0.536 (0.962)
  Streaming, 6 months: number analyzed (Participants) | 27
  Streaming, 6 months | 0.444 (0.698)

27. Secondary Outcome: Usability Information: Battery Lifetime of Sound Processor
Description: Average hours of battery lifetime
Time Frame: At 6 weeks, 3 months and 6 months after surgery
Population: For some participants the data are not available at all visits.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
hours
  6 weeks: number analyzed (Participants) | 27
  6 weeks | 27.3 (15.0)
  3 months | 27.4 (11.2)
  6 months: number analyzed (Participants) | 26
  6 months | 24.3 (12.4)

28. Secondary Outcome: Difference in Hearing Performance Between the Osia 2 System and a Baha 5 Power Sound Processor on a Baha Softband (Preoperative) at 4 Weeks, 3 Months and 6 Months Post Surgery Assessed Via Audiometric Thresholds
Description: Free-field [Pure Tone Average (PTA) 4, Mean of 0.5, 1, 2 and 4 kHz].
Time Frame: Baseline before surgery, 4 weeks, 3 months and 6 months after surgery
Population: Some participants did not perform the test at all visits.
Measure: Mean (Standard Deviation); unit: db HL (decibel Hearing Level)
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
db HL (decibel Hearing Level)
  PTA4, 4 weeks: number analyzed (Participants) | 27
  PTA4, 4 weeks | 0.046 (7.134)
  PTA4, 3 months: number analyzed (Participants) | 27
  PTA4, 3 months | -1.62 (6.41)
  PTA4, 6 months | -2.54 (8.32)

29. Secondary Outcome: Difference in Hearing Performance Between the Osia 2 System and a Baha 5 Power Sound Processor on a Baha Softband (Preoperative) at 4 Weeks, 3 Months and 6 Months Post Surgery Assessed Via Audiometric Thresholds
Description: Free-field [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 and 8.0 kHz].
Time Frame: Baseline before surgery, 4 weeks, 3 months and 6 months after surgery
Population: Some participants did not perform the test at all visits.
Measure: Mean (Standard Deviation); unit: db HL (decibel Hearing Level)
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
db HL (decibel Hearing Level)
  0.25 kHz, 4 weeks: number analyzed (Participants) | 27
  0.25 kHz, 4 weeks | 4.44 (13.18)
  0.5 kHz, 4 weeks: number analyzed (Participants) | 27
  0.5 kHz, 4 weeks | 4.44 (10.13)
  0.75 kHz, 4 weeks: number analyzed (Participants) | 27
  0.75 kHz, 4 weeks | -0.741 (6.893)
  1.0 kHz, 4 weeks: number analyzed (Participants) | 27
  1.0 kHz, 4 weeks | 1.85 (7.61)
  1.5 kHz, 4 weeks: number analyzed (Participants) | 27
  1.5 kHz, 4 weeks | 0.185 (8.376)
  2.0 kHz, 4 weeks: number analyzed (Participants) | 27
  2.0 kHz, 4 weeks | -2.22 (8.70)
  3.0 kHz, 4 weeks: number analyzed (Participants) | 27
  3.0 kHz, 4 weeks | -1.48 (10.27)
  4.0 kHz, 4 weeks: number analyzed (Participants) | 27
  4.0 kHz, 4 weeks | -3.89 (11.21)
  6.0 kHz, 4 weeks: number analyzed (Participants) | 27
  6.0 kHz, 4 weeks | -11.9 (10.9)
  8.0 kHz, 4 weeks: number analyzed (Participants) | 27
  8.0 kHz, 4 weeks | 4.78 (16.49)
  0.25 kHz, 3 months: number analyzed (Participants) | 27
  0.25 kHz, 3 months | 3.15 (10.57)
  0.5 kHz, 3 months: number analyzed (Participants) | 27
  0.5 kHz, 3 months | 3.15 (9.11)
  0.75 kHz, 3 months: number analyzed (Participants) | 27
  0.75 kHz, 3 months | -2.59 (6.70)
  1.0 kHz, 3 months: number analyzed (Participants) | 27
  1.0 kHz, 3 months | 1.11 (6.55)
  1.5 kHz, 3 months: number analyzed (Participants) | 27
  1.5 kHz, 3 months | -0,370 (7,836)
  2.0 kHz, 3 months: number analyzed (Participants) | 27
  2.0 kHz, 3 months | -3.52 (8.64)
  3.0 kHz, 3 months: number analyzed (Participants) | 27
  3.0 kHz, 3 months | -1.85 (10.48)
  4.0 kHz, 3 months: number analyzed (Participants) | 27
  4.0 kHz, 3 months | -7.22 (10.41)
  6.0 kHz, 3 months: number analyzed (Participants) | 27
  6.0 kHz, 3 months | -13.3 (10.3)
  8.0 kHz, 3 months: number analyzed (Participants) | 27
  8.0 kHz, 3 months | 1.63 (15.20)
  0.25 kHz, 6 months | 3.93 (13.77)
  0.5 kHz, 6 months | 2.86 (9.95)
  0.75 kHz, 6 months | -2.68 (8.76)
  1.0 kHz, 6 months | -1.07 (7.98)
  1.5 kHz, 6 months | -3.39 (7.34)
  2.0 kHz, 6 months | -4.64 (10.97)
  3.0 kHz, 6 months | -3.04 (12.35)
  4.0 kHz, 6 months | -7.32 (11.26)
  6.0 kHz, 6 months | -13.9 (13.6)
  8.0 kHz, 6 months | 2.86 (17.87)

30. Secondary Outcome: Difference in Hearing Performance Between the Osia 2 System and a Baha 5 Power Sound Processor on a Baha Softband (Preoperative) at 4 Weeks, 3 Months and 6 Months Post Surgery Assessed Via Adaptive Speech Recognition in Noise
Description: Signal-to-noise ratio, 50% speech understanding
Time Frame: Baseline before surgery, 4 weeks, 3 months and 6 months after surgery
Population: Some participants did not perform the test at all visits.
Measure: Mean (Standard Deviation); unit: db SNR (decibel Speech in Noise Ratio)
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
db SNR (decibel Speech in Noise Ratio)
  4 weeks: number analyzed (Participants) | 27
  4 weeks | -0.870 (1.366)
  3 months: number analyzed (Participants) | 27
  3 months | -1.21 (1.42)
  6 months | -0.846 (1.587)

31. Secondary Outcome: Difference in Hearing Performance Between the Osia 2 System and a Baha 5 Power Sound Processor on a Baha Softband (Preoperative) at 4 Weeks, 3 Months and 6 Months Post Surgery Assessed Via Speech Recognition in Quiet
Description: % correctly perceived words at 50dB, 65dB and 80dB SPL
Time Frame: Baseline before surgery, 4 weeks, 3 months and 6 months after surgery
Population: Some participants did not perform all tests at all visits.
Measure: Mean (Standard Deviation); unit: Percentage of correct words
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
Percentage of correct words
  Speech in quiet at 50 dB, 4 weeks: number analyzed (Participants) | 27
  Speech in quiet at 50 dB, 4 weeks | 12.2 (18.3)
  Speech in quiet at 65 dB, 4 weeks: number analyzed (Participants) | 27
  Speech in quiet at 65 dB, 4 weeks | 9.77 (14.76)
  Speech in quiet at 80 dB, 4 weeks: number analyzed (Participants) | 27
  Speech in quiet at 80 dB, 4 weeks | 2.88 (10.21)
  Speech in quiet at 50 dB, 3 months: number analyzed (Participants) | 27
  Speech in quiet at 50 dB, 3 months | 13.2 (18.8)
  Speech in quiet at 65 dB, 3 months: number analyzed (Participants) | 27
  Speech in quiet at 65 dB, 3 months | 10.1 (16.0)
  Speech in quiet at 80 dB, 3 months: number analyzed (Participants) | 27
  Speech in quiet at 80 dB, 3 months | 2.66 (10.13)
  Speech in quiet at 50 dB, 6 months | 10.7 (18.3)
  Speech in quiet at 65 dB, 6 months | 8.84 (15.22)
  Speech in quiet at 80 dB, 6 months | 4.00 (8.26)

32. Secondary Outcome: Hearing Performance Using a Baha Softband (Preoperative) at Baseline and the Osia 2 System at 4 Weeks, 3 Months and 6 Months Post Surgery Assessed Via Bone Conduction (BC) Direct
Description: BC direct (0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0 and 6.0 kHz)
Time Frame: Baseline before surgery, 4 weeks, 3 months and 6 months after surgery
Population: Some participants did not perform the test at all visits.
Measure: Mean (Standard Deviation); unit: db HL (decibel Hearing Level)
Arm/Group | Osia 2 System
Number analyzed (Participants) | 28
db HL (decibel Hearing Level)
  BC Direct 250 Hz, baseline | 13.2 (10.2)
  BC Direct 500 Hz, baseline | 24.7 (11.3)
  BC Direct 750 Hz, baseline | 20.7 (12.4)
  BC Direct 1000 Hz, baseline | 20.0 (13.5)
  BC Direct 1500 Hz, baseline | 19.1 (14.6)
  BC Direct 2000 Hz, baseline | 31.2 (15.3)
  BC Direct 3000 Hz, baseline | 36.8 (18.7)
  BC Direct 4000 Hz, baseline | 43.5 (17.6)
  BC Direct 6000 Hz, baseline | 46.1 (17.6)
  BC Direct 250 Hz, 4 weeks | 5.18 (12.87)
  BC Direct 500 Hz, 4 weeks | 14.5 (8.7)
  BC Direct 750 Hz, 4 weeks | 5.71 (11.20)
  BC Direct 1000 Hz, 4 weeks | 9.46 (11.33)
  BC Direct 1500 Hz, 4 weeks | 7.50 (13.23)
  BC Direct 2000 Hz, 4 weeks | 12.0 (14.2)
  BC Direct 3000 Hz, 4 weeks | 13.9 (15.4)
  BC Direct 4000 Hz, 4 weeks | 23.8 (17.1)
  BC Direct 6000 Hz, 4 weeks | 22.0 (18.7)
  BC Direct 250 Hz, 3 months: number analyzed (Participants) | 15
  BC Direct 250 Hz, 3 months | 4.00 (11.21)
  BC Direct 500 Hz, 3 months: number analyzed (Participants) | 15
  BC Direct 500 Hz, 3 months | 13.0 (9.8)
  BC Direct 750 Hz, 3 months: number analyzed (Participants) | 15
  BC Direct 750 Hz, 3 months | 4.33 (12.08)
  BC Direct 1000 Hz, 3 months: number analyzed (Participants) | 15
  BC Direct 1000 Hz, 3 months | 9.67 (13.29)
  BC Direct 1500 Hz, 3 months: number analyzed (Participants) | 15
  BC Direct 1500 Hz, 3 months | 6.67 (15.43)
  BC Direct 2000 Hz, 3 months: number analyzed (Participants) | 15
  BC Direct 2000 Hz, 3 months | 14.0 (15.9)
  BC Direct 3000 Hz, 3 months: number analyzed (Participants) | 15
  BC Direct 3000 Hz, 3 months | 13.3 (18.5)
  BC Direct 4000 Hz, 3 months: number analyzed (Participants) | 15
  BC Direct 4000 Hz, 3 months | 24.3 (17.4)
  BC Direct 6000 Hz, 3 months: number analyzed (Participants) | 15
  BC Direct 6000 Hz, 3 months | 27.0 (18.5)
  BC Direct 250 Hz, 6 months: number analyzed (Participants) | 21
  BC Direct 250 Hz, 6 months | 8.10 (13.83)
  BC Direct 500 Hz, 6 months: number analyzed (Participants) | 21
  BC Direct 500 Hz, 6 months | 15.0 (8.5)
  BC Direct 750 Hz, 6 months: number analyzed (Participants) | 21
  BC Direct 750 Hz, 6 months | 6.90 (12.60)
  BC Direct 1000 Hz, 6 months: number analyzed (Participants) | 21
  BC Direct 1000 Hz, 6 months | 10.7 (11.3)
  BC Direct 1500 Hz, 6 months: number analyzed (Participants) | 21
  BC Direct 1500 Hz, 6 months | 5.95 (13.84)
  BC Direct 2000 Hz, 6 months: number analyzed (Participants) | 21
  BC Direct 2000 Hz, 6 months | 14.3 (13.7)
  BC Direct 3000 Hz, 6 months: number analyzed (Participants) | 21
  BC Direct 3000 Hz, 6 months | 13.6 (17.0)
  BC Direct 4000 Hz, 6 months: number analyzed (Participants) | 21
  BC Direct 4000 Hz, 6 months | 25.7 (16.9)
  BC Direct 6000 Hz, 6 months: number analyzed (Participants) | 21
  BC Direct 6000 Hz, 6 months | 25.0 (18.8)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events are presented by the CTCAE term.
Arm/Group | Osia 2 System
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 3/29
Other Adverse Events (participants affected / at risk) | 21/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osia 2 System (N=29)
Gastroenteritis (Infections and infestations) | 1 (29)
Infected Skin/ Wound With Subcutaneous Collection (Infections and infestations) | 1 (29)
Infected Wound/Possible Flap Compromise (Infections and infestations) | 1 (29)
Preoperative Bradycardia (Cardiac disorders) | 1 (29)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osia 2 System (N=29)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 5 (29)
General disorders and administration site conditions - Other (General disorders) | 5 (29)
Wound infection (Infections and infestations) | 4 (29)
Wound complication (Injury, poisoning and procedural complications) | 6 (29)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (29)
Psychiatric Disorders - Other (Psychiatric disorders) | 2 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institutions agree that no publication of the study results may be made until publication of the results of the multi-centre study or 2 years after study completion, whichever is the sooner.

DOCUMENTS (2):
  • Study Protocol (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT04041700/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT04041700/SAP_001.pdf